CLINICAL TRIAL: NCT05102747
Title: Stereotactic Radiotherapy in Oligometastatic Brain Disease: a Randomised Phase III Study Comparing Hypofractionated Stereotactic Radiation Therapy (3*10 Gy) to the Historical Single-dose Radiosurgery (1*20 to 25 Gy) With Medico-economic Evaluation.
Acronym: OligoBM-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: Association de Neuro-Oncologues d'Expression Francaise (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-A01622-39
Record Dates: First submitted 2021-10-06; First posted 2021-11-01 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Brain Metastasis; Oligoprogression
Keywords: Stereotactic radiosurgery; Fractionated stereotactic radiotherapy
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery; Health Records, Personal; Spermine Synthase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated SRT (stereotactic radiotherapy) (Experimental)
  Interventions: Radiation: Hypofractionated SRT (stereotactic radiotherapy)
- Historical single-dose SRS (stereotactic radiosurgery) (Active Comparator)
  Interventions: Radiation: Historical single-dose SRS (stereotactic radiosurgery)

INTERVENTIONS:
Radiation: Hypofractionated SRT (stereotactic radiotherapy) — 3*10Gy over 1 week
  Arms: Hypofractionated SRT (stereotactic radiotherapy)
Radiation: Historical single-dose SRS (stereotactic radiosurgery) — 20 to 25Gy/1 fraction
  Arms: Historical single-dose SRS (stereotactic radiosurgery)

SUMMARY:
Brain metastases (BM) are a common systemic cancer manifestation which incidence increases. Therapeutic options include whole-brain radiotherapy (WBRT), surgery, and stereotactic radiosurgery (SRS). The concept of "oligometastatic" cerebral disease (oligoBM) has emerged and led to consider alternative approaches. The main challenge is to preserve neurological function and independence the longest as possible.

Stereotactic radiotherapy (SRT) has emerged as an alternative treatment modality for selected oligoBM patients. It allows to achieve the balance of tumour destruction and normal tissue preservation by precisely and accurately delivering a very high dose of radiation in one (SRS) or a few (HSRT) fractions to a limited, well-defined volume. However, no standard exists for decision-making between SRS and HSRT and this important question is being discussed in the recent literature.

HSRT appears particularly interesting, assuming the patient convenience of few fractions, the normal tissue sparing achieved through focal irradiation, and the improved normal tissue tolerance of high dose radiation through fractionation.

Common adverse effects of SRT are rare but can occasionally be serious, notably radionecrosis that may induce neurological deficits in patients. Although SRS is often less well-tolerated, it remains the mainstay of treatment.

To investigators knowledge, SRS and HSRT have not been prospectively compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* WHO performance status 0 or 1;
* Patient eligible for SRT after a multidisciplinary committee decision; Patient with BMs from radioresistant cancer (renal cell carcinoma, sarcoma, melanoma) is eligible
* Patient having up to 5 BM of solid tumours with an histologically proven diagnoses; patients who have had a metastasectomy and having 1 to 4 BM lesions is eligible (ANOCEF recommendations); post-operative cavity must be treated by radiosurgery according to local procedures with respect of non-inclusion criteria* (cavity will not be analyzed for efficacy)
* Presence of at least one and no more than 5 target lesions for SRT, measuring between 10 and 25 mm. In the event of synchronous BM, lesions measuring less than 10mm or more than 25mm (1 to 4 lesions) will be treated at the discretion of the investigator
* Max cumulative GTV of 30cm3
* Normal complete blood count (CBC)
* Absence of bleeding BM or meningeal carcinomatosis;
* Symptomatic BM are allowed
* DS-GPA score:

  * Renal cancer: DS-GPA 2,5 or more
  * Breast cancer: DS-GPA 2,5 or more
  * Melanoma: DS-GPA 1.5 or more
  * Gastro-instestinal (GI) cancer: DSGPA 3 or more
  * Adenocarcinoma lung cancer: DS-GPA 2 or more (DS-GPAmol)
  * Squamous lung cancer : DS-GPA 2,5 or more (DS-GPAmol)
  * For cancers where the DS-GPA score is not applicable, the patient is eligible if eligibility criteria are met
* Patient with no concomitant systemic treatment; in case of ongoing systemic treatment, wash out period of 3-7 days before and after SRT, depending of drug and at the discretion of investigator;
* Patient sufficiently cooperating to perform the treatment with the use of a thermoformed mask;
* Patient whose neuropsychological abilities allow to follow the requirements of the protocol;
* Female with childbearing potential must use adequate contraception
* Signed informed consent formOligoBM-01 Trial - ID-RCB number: 2021-A01622-39 - version 3.1 dated from 2023-06-22 Page 9 of 51
* Patients affiliated to the social security system

Exclusion Criteria:

* Patients with current or past history small cell lung cancer, germ-cell tumours, lymphoma, leukemia and multiple myeloma within the last 5 years;
* Patients with metastases in the brain stem, or within 1 cm of the optic apparatus;
* Patients with an associated neurodegenerative disease;
* Any symptoms not attributable to BM or cancer disease requiring long term corticosteroid use (regardless of dose);
* Contraindication to perform the brain MRI or gadolinium or iodinated contrast;
* Known hypersensitivity to the contrast product or to any their excipients
* Patients with previous brain stereotactic irradiation
* Whole brain irradiation history;
* Haemorrhagic metastasis;
* Ongoing anti angiogenic treatment (treatment should be held 3-7 days before irradiation and re-initiated 3-7 days after irradiation for patient to be eligible);
* Patients with too close brain lesions for whom a treatment plan on one target metastasis delivers a dose > 5 Gy on other concomitant metastasis ;
* Patient deprived of liberty or under guardianship;
* Known pregnancy or breastfeeding
* Any geographical conditions, social and associated psychopathology that may compromise the patient's ability to participate in the study;
* Participation in a therapeutic trial for less than 30 days.
* Patient deprived of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2023-01-12 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Local control assessed by RANO-BM criteria | 12 months

SECONDARY OUTCOMES:
Brain acute and late toxicities assessed by NCI CTCAE v5.0 | 12 months
Radionecrosis by RANO-BM criteria | 12 months

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHU, Bordeaux
  - Institut Bergonié, Bordeaux
  - CHU, Brest
  - Centre François Baclesse, Caen
  - CHU, Grenoble
  - Centre Guillaume le Conquérant, Le Havre
  - Groupe hospitalier Bretagne Sud, Lorient
  - Centre Antoine Lacassagne, Nice
  - La Pitié Salpétrière, Paris
  - Centre hospitalier Lyon Sud, Pierre-Bénite
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre d'Oncologie et Radiothérapie Saint-Jean, Saint-Doulchard
  - Institut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif